CLINICAL TRIAL: NCT00117806
Title: A Spinal Cord Injury Vocational Integration Program: Implementation and Outcomes
Brief Title: Spinal Cord Injury Vocational Integration Program (SCI-VIP)
Acronym: SCI-VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3773-R
Record Dates: First submitted 2005-07-01; First posted 2005-07-08 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injuries
Keywords: Adult; Depression; Employment, supported; Health Service/ut; Humans; Outcomes; Quality of life; Veterans/rh (rehabilitation); Workplace; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries; Depression | interventions — DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): SCI-VIP: Supported employment implemented for veterans with spinal cord injury
  Interventions: Behavioral: Arm 1
- Arm 2 (Placebo Comparator): Standard Care: varies slightly between participating VA SCI centers, however, usually involves referral outside SCI center
  Interventions: Behavioral: Arm 2

INTERVENTIONS:
Behavioral: Arm 1 — SCI-VIP: Supported employment implemented for veterans with spinal cord injury.
  Arms: Arm 1
Behavioral: Arm 2 — Standard Care: varies slightly between participating VA SCI centers, however, usually involves referral outside SCI center
  Arms: Arm 2

SUMMARY:
This study involves research about how to help Veterans with spinal cord injury (SCI) gain employment. During the first couple of years following SCI, many people are concentrating on their rehabilitation and are unable to afford the time for return to work. However, studies have shown people often regain the necessary strength and function about two years after SCI to resume activities of daily living very similar to what they experienced prior to the SCI. Even though many social and legal efforts have been made in the last decade to improve chances for people with disabilities to return to work, Veterans with SCI are sometimes hindered in finding employment because of age, past work history, and many other factors. Other Veterans with SCI are very successful at finding employment either working for themselves or working for a company. The investigators know very little about what issues Veterans with SCI face when they attempt to find employment after SCI. The study will analyze both quantitative and qualitative measures to maximize its findings.

DETAILED DESCRIPTION:
Legal mandates, such as the Rehabilitation Act of 1973 and the Americans with Disabilities Act, have been implemented to improve employment opportunities for disabled persons and yet the proportion of persons with spinal cord injury (SCI) who are employed remains about 9%. For the Veteran population with SCI, the return to work rate is most likely much lower. This study will be conducted to evaluate whether a vocational rehabilitation program patterned after the VA Community Employment and Support approach improves rehabilitation outcomes for the SCI Veteran population as compared with vocational rehabilitation practices currently used in most Veteran Affairs Medical Centers (VAMCs). The vocational rehabilitation program developed for the SCI Veterans is referred to as SCI-VIP and it will be implemented at the Dallas VA Medical Center (VAMC), Houston VAMC, San Diego VAMC, and Cleveland VAMC. A five year evaluative research will be conducted to test the following hypothesized outcomes (HO) from the subjects who participate in the SCI-VIP program and a control group of subjects who receive conventional methods of vocational rehabilitation:

Primary HO: Veterans with SCI who participate in the SCI-VIP will demonstrate significantly greater changes in vocational rehabilitation after twelve months than those who do not receive this intervention. Vocational rehabilitation will be a measure of change from baseline to one-year in the subject's scores on instruments which measure employment indices, perceived barriers to employment, level of handicap, quality of life, depression, and sustaining care needs.

Secondary HO 1: Veterans with SCI who participate in the SCI-VIP will exhibit lower VA and non-VA costs for medical, non-rehabilitation treatment, offsetting the higher SCI-VIP program costs.

Secondary HO 2: The program fidelity will be equally adequate in terms of accomplishing program objectives relative to operations, cost-benefit balance, subject and stakeholder satisfaction, and outcomes when comparing the four SCI-VIP programs and when comparing conventional vocational rehabilitation approaches applied at six different VAMCs.

Program evaluation and cost-benefit analysis will be conducted using a fidelity instrument developed by the researchers and patterned after fidelity instruments conventionally used to evaluate psychiatric rehabilitation programs. Veterans at each VAMC who express an interest in vocational rehabilitation and consent to participate in this study will be randomized to either the experimental or the control group. It is expected that at least 96 subjects will participate in the SCI-VIP approach to vocational rehabilitation and 144 Veterans who receive conventional vocational rehabilitation will form the control group.

Data will be collected from subjects upon enrollment into either the experimental or control group and every three months for one year. Descriptive analysis will be used to compare differences between groups of subjects drawn from each VAMC and to compare participants in the experimental and control groups. Analysis of variance will be computed to determine degree of difference between experimental group and control group subjects' scores on each dependent variable. The study hypotheses will be tested using the Mann-Whitney U, Chi-square, and odds ratio statistical procedures. The Cochran-Mantel-Haenszel along with relative risk scores will indicate the likelihood that any change in performance between baseline and program completion for ether experimental or control group subjects could be attributed to the subjects' degree of participation in the SCI-VIP, which VAMC vocational rehabilitation services were received, SCI factors, and age.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years old - Spinal cord injured as a result of trauma or disease
* Medically and neurologically stable
* Lives within the metropolitan area that is proximal to the VAMC (Cleveland, Dallas, Houston, San Diego, St. Louis)
* Has access to transportation
* Expresses an interest in competitive employment as an outcome of participation
* Willingly signs a consent form indicating voluntary and informed participation in the study

Exclusion Criteria:

* Medically and/or surgically unstable
* Unwilling to complete the consenting process
* Mentally impaired such that independent reasoning and judgment jeopardize safety of self and others
* Currently involved in untreated alcohol and/or drug dependency
* Employed in a compensated job at the time of recruitment and earning above SGA ($940/month in 2008) - Lives more than approximately 100 miles from the participating VAMC SCI Center

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ottomanelli, PhD, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (5):
- United States (5):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - VA Medical Center, St Louis, St Louis, Missouri
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas

REFERENCES:
- [Background] Ottomanelli L, Goetz LL, McGeough C, Kashner TM. Building research capacity through partnerships: Spinal Cord Injury-Vocational Integration Program Implementations and Outcomes inaugural meeting. J Rehabil Res Dev. 2007;44(1):vii-xii. doi: 10.1682/jrrd.2006.06.0072. No abstract available. PMID 17551852
- [Background] Ottomanelli L, Lind L. Review of critical factors related to employment after spinal cord injury: implications for research and vocational services. J Spinal Cord Med. 2009;32(5):503-31. doi: 10.1080/10790268.2009.11754553. PMID 20025147
- [Background] Ottomanelli L, Goetz L, McGeough C, Suris A, Sippel J, Sinnott P, Wagner TH, Cipher DJ. Methods of a multisite randomized clinical trial of supported employment among veterans with spinal cord injury. J Rehabil Res Dev. 2009;46(7):919-30. doi: 10.1682/jrrd.2008.10.0145. PMID 20104414
- [Background] Thomas FP, Goetz LL, Dixon T, Ho C, Holmes SA, Sandford P, Smith S, Ottomanelli L. Optimizing medical care to facilitate and sustain employment after spinal cord injury. J Rehabil Res Dev. 2014;51(6):xi-xxii. doi: 10.1682/JRRD.2014.05.0119. No abstract available. PMID 25479192
- [Result] Ottomanelli L, Goetz LL, Suris A, McGeough C, Sinnott PL, Toscano R, Barnett SD, Cipher DJ, Lind LM, Dixon TM, Holmes SA, Kerrigan AJ, Thomas FP. Effectiveness of supported employment for veterans with spinal cord injuries: results from a randomized multisite study. Arch Phys Med Rehabil. 2012 May;93(5):740-7. doi: 10.1016/j.apmr.2012.01.002. PMID 22541306
- [Result] Ottomanelli L, Barnett SD, Goetz LL. A prospective examination of the impact of a supported employment program and employment on health-related quality of life, handicap, and disability among Veterans with SCI. Qual Life Res. 2013 Oct;22(8):2133-41. doi: 10.1007/s11136-013-0353-5. Epub 2013 Jan 24. PMID 23345022
- [Result] Ottomanelli L, Barnett SD, Goetz LL. Effectiveness of supported employment for veterans with spinal cord injury: 2-year results. Arch Phys Med Rehabil. 2014 Apr;95(4):784-90. doi: 10.1016/j.apmr.2013.11.012. Epub 2013 Dec 4. PMID 24316325
- [Result] Sinnott PL, Joyce V, Su P, Ottomanelli L, Goetz LL, Wagner TH. Cost-effectiveness of supported employment for veterans with spinal cord injuries. Arch Phys Med Rehabil. 2014 Jul;95(7):1254-61. doi: 10.1016/j.apmr.2014.01.010. Epub 2014 Jan 31. PMID 24486426
- [Result] Smith-Morris C, Lopez G, Ottomanelli L, Goetz L, Dixon-Lawson K. Ethnography, fidelity, and the evidence that anthropology adds: supplementing the fidelity process in a clinical trial of supported employment. Med Anthropol Q. 2014 Jun;28(2):141-61. doi: 10.1111/maq.12093. Epub 2014 Apr 21. PMID 24752942
- [Result] Ottomanelli L, Barnett SD, Toscano R. Individual placement and support (IPS) in physical rehabilitation and medicine: the VA spinal cord injury experience. Psychiatr Rehabil J. 2014 Jun;37(2):110-2. doi: 10.1037/prj0000079. PMID 24912059
- [Result] LePage J, Ottomanelli L, Barnett SD, Njoh EN. Spinal cord injury combined with felony history: effect on supported employment for Veterans. J Rehabil Res Dev. 2014;51(10):1497-504. doi: 10.1682/JRRD.2014.02.0045. PMID 25856266
- [Result] Ottomanelli L, Barnett SD, Goetz LL, Toscano R. Vocational rehabilitation in spinal cord injury: what vocational service activities are associated with employment program outcome? Top Spinal Cord Inj Rehabil. 2015 Winter;21(1):31-9. doi: 10.1310/sci2101-31. PMID 25762858

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two-hundred forty-nine subjects were enrolled in the study which, 48 were excluded for various reasons including benefits (n=19), age >65 (n=10), currently employed (n=6), and other (n=13), leaving 201 subjects. For the purposes of reporting the 44 veterans in the observational site were not included, therefore there are only 157 subjects included.
Groups:
- Supported Employment: SCI-VIP: evidence-based supported employment implemented for veterans with spinal cord injury
  Evidence-Based Supported Employment Vocational Rehabilitation: SCI-VIP: evidence-based supported employment implemented for veterans with spinal cord injury.
- Treatment As Usual: Standard Care: varies slightly between participating VA SCI centers, however, usually involves referral outside SCI center
Period: Overall Study
Arm/Group | Supported Employment | Treatment As Usual
Started | 81 | 76
Completed | 43 | 60
Not Completed | 38 | 16

BASELINE CHARACTERISTICS:
Population: AIS DATA-Missing 1 participant for Supported Employment and Treatment As Usual groups.
  AIS & Neurologival Level- Missing 1 participant for Supported employment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Supported Employment | Treatment As Usual | Total
Number analyzed (Participants) | 81 | 76 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 76 | 157
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (9.8) | 49.8 (9.8) | 49.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 77 | 72 | 149
Race/Ethnicity, Customized [Number; unit: participants]
  White | 37 | 33 | 70
  African American | 29 | 37 | 66
  Hispanic | 5 | 1 | 6
  Other | 10 | 5 | 15
Functional Independence Measure [Mean (Standard Deviation); unit: units on a scale] — The FIM is an 18-item instrument that assesses disability in terms of what level of assistance an individual needs to perform various activities. Each item is on a scale from 1 (total assistance) to 7 (complete independence). Motor subscale scores range from 13 (total dependence) to 91 (total independence) and cognitive subscale scores range from 5 (total dependence) to 35 (total independence). Motor and Cognitive are summed to create the Total FIM scores which range from 18 (totally dependent) to 126 (totally independent).
  units on a scale
    Total | 98.9 (23.8) | 98.2 (23.7) | 98.6 (23.6)
    Cognitive | 33.8 (2.3) | 33.7 (2.8) | 33.8 (2.5)
    Motor | 66.9 (21.6) | 66.4 (22.2) | 66.6 (21.8)
Measures of Handicap (CHART) [Mean (Standard Deviation); unit: units on a scale] — The CHART contains 32 items assessing six dimensions of a person's handicap: cognitive independence, physical independence, mobility, occupation, social integration, and economic self-sufficiency. A minimum score of 0 indicating full handicap in an individual's ability to sustain an individual existence and maximum score of 100 indicating no handicap in an individual's ability to sustain an individual existence , is permitted for each subscale.
  units on a scale
    Social Integration | 82.0 (13.6) | 84.7 (12.7) | 83.3 (13.1)
    Mobility | 80.4 (17.0) | 80.4 (22.4) | 80.4 (19.7)
    Cognitive | 89.4 (16.6) | 90.8 (14.9) | 90.1 (15.7)
    Occupation | 51.5 (32.9) | 50.4 (30.6) | 51.0 (31.7)
    Physical | 85.7 (20.9) | 87.2 (22.1) | 86.4 (21.4)
    Economic Self Sufficiency | 51.5 (37.8) | 52.6 (36.9) | 52.1 (15.7)
Quality of Life VR-36 [Mean (Standard Deviation); unit: units on a scale] — The VR-36 is a 36-item instrument which assesses general health-related quality of life. The VR-36 assesses eight domains of a person's health and functioning: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. The item responses are on a 3-point scale ranging from "Yes, limited a lot" to "No, not limited at all." The items are summed and the range is from 0-100, 100 is equivalent to maximum health.
  units on a scale
    Mental Component Score | 54.7 (13.8) | 55.6 (12.9) | 55.1 (13.3)
    Physical Component Score | 27.7 (7.5) | 28.1 (8.4) | 27.9 (7.9)
ASIA Impairment Scale (AIS) [Number; unit: participants] — The ASIA Impairment Scale is a tool used to categorize motor & sensory impairment in individuals with SCI. A-Comp B-Incomp: Sensory but not motor function is preserved below the neurological level & includes the sacral segments S4-S5. C-Incomplete: Motor function is preserved below the neuro level & more than half of key muscles below the neuro level have a muscle grade < 3. D-Incomplete: Motor function is preserved below the neuro level, and at least half of key muscles below the neuro level have a muscle grade of >=3; E-Normal.
  Data were not available for all participants. Incomplete data.
  participants
    A-Complete | 26 | 20 | 46
    B-Sensory Incomplete | 11 | 13 | 24
    C-Motor Incomplete | 18 | 18 | 36
    D-Motor Incomplete | 25 | 21 | 46
    E-Normal | 0 | 4 | 4
AIS and neurological Level [Number; unit: participants] — Data were not available for all participants.
  participants
    High tetraplegia, AIS A, B,C | 12 | 13 | 25
    Low tetraplegia, AIS A, B, C | 5 | 10 | 15
    Paraplegia, AIS A, B, C | 38 | 27 | 65
    AIS D/E | 25 | 25 | 50
Marital Status [Number; unit: participants]
  Married | 30 | 15 | 45
  Divorced | 28 | 34 | 62
  Other | 23 | 27 | 50
Education Years [Mean (Standard Deviation); unit: years] | 13.1 (2.3) | 13.5 (1.9) | 13.3 (2.2)
VA benefits recipient [Number; unit: participants] — Data were not available for all participants. Not all veterans were recipients of VA benefits.
  participants | 50 | 43 | 93
Service-connected benefits for SCI recipient [Number; unit: participants] — Data were not available for all participants. Not all veterans received service-connected benefits.
  participants | 19 | 15 | 34
Service-connected 100% [Number; unit: participants] — Data were not available for all participants. Not all veterans were 100% service-connected.
  participants | 16 | 13 | 29
No Service-connected/Non-service-connected benefits [Number; unit: participants] — Data were not available for all participants. Not all veterans received service-connected or non-service connected benefits.
  participants | 26 | 20 | 46
Non-service-connected pension [Number; unit: participants] — Data were not available for all participants. Not all veterans received non-service-connected benefits.
  participants | 18 | 18 | 36
Monthly non-service-connected amount [Mean (Standard Deviation); unit: dollars] | 1024 (482) | 986 (421) | 1005.7 (447.9)
Social Security Income recipient [Number; unit: participants] — Data were not available for all participants. Not all veterans received SSI.
  participants | 10 | 11 | 21
Social Security Disability Insurance recipient [Number; unit: participants] — Data were not available for all participants. Not all veterans were recipients of SSDI.
  participants | 45 | 46 | 91
Neither Social Security Income/Social Security Disability Insurance recipient [Number; unit: participants] — Data were not available for all participants. Some veterans were neither recipients of SSI & SSDI.
  participants | 26 | 20 | 46

OUTCOME MEASURES:

1. Primary Outcome: Competitive Employment-Total Jobs
Description: Competitive employment (a job in the community paying minimum wage ) during year 1 among those subjects obtaining employment.
Time Frame: 12 months
Measure: Number; unit: Total Competitive Employments
Groups:
- Supported Employment: Supported Employment Vocational Rehabilitation: SCI-VIP: supported employment implemented for veterans with spinal cord injury.
Arm/Group | Supported Employment | Treatment As Usual
Number analyzed (Participants) | 81 | 76
Total Competitive Employments | 50 | 21

2. Primary Outcome: Competitive Employment-Participants With Competitive Employment
Description: as for outcome 1
Time Frame: 12 months
Measure: Number; unit: Participants with competitive employment
Arm/Group | Supported Employment | Treatment As Usual
Number analyzed (Participants) | 81 | 76
Participants with competitive employment | 21 | 8

3. Primary Outcome: Competitive Employment-Percentage of Participants With Competitive Employment
Description: Employment outcomes during year 1 among those subjects obtaining competitive employment.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm 1: SCI-VIP: evidence-based supported employment implemented for veterans with spinal cord injury
  Evidence-Based Supported Employment Vocational Rehabilitation: SCI-VIP: evidence-based supported employment implemented for veterans with spinal cord injury.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 81 | 76
percentage of participants | 25.9 [17.6 to 36.5] | 10.5 [3.6 to 17.4]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority or Other; p = 0.008, Chi-squared

ADVERSE EVENTS:
Description: Within the required number of days (per IRB) of becoming aware of any local unanticipated SAE in VA research, members of the VA research community are required to ensure that the SAE has been reported in writing to the IRB.This is in addition to other reporting requirements.Finally an annual report of SAEs is reviewed by data monitoring committee.
Groups:
- Supported Employment: SCI-VIP: supported employment implemented for veterans with spinal cord injury
  Supported Employment Vocational Rehabilitation: SCI-VIP: supported employment implemented for veterans with spinal cord injury.
Arm/Group | Supported Employment | Treatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/76
Other Adverse Events (participants affected / at risk) | 0/81 | 0/76

LIMITATIONS AND CAVEATS:
Majority of sample is male; Potential selection bias (participants who decided to remain in study for second year may be different from those who did not though no statistical significance was detected between groups)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No